CLINICAL TRIAL: NCT01112410
Title: A Randomised Double Blind 13 Week Crossover Trial of Hypertonic Saline (6%) Versus Isotonic Saline (0.9%) in Patients With Bronchiectasis.
Brief Title: Hypertonic Saline (6%) Versus Isotonic Saline (0.9%) in Bronchiectasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Belfast Health and Social Care Trust (Other)
Responsible Party: Dr Judy Bradley, Belfast Health and Social Care Trust
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 09023JB-OPMS
Record Dates: First submitted 2010-04-27; First posted 2010-04-28 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-01

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Hypertonic saline
MeSH Terms: conditions — Bronchiectasis | interventions — Saline Solution, Hypertonic; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Hypertonic saline — Hypertonic saline (6%) nebulised twice a day for 4 weeks.
  (Randomised crossover trial)
Other: Isotonic saline — Isotonic Saline (0.9%) nebulised twice a day for 4 weeks.

SUMMARY:
The investigators hypothesise that nebulised hypertonic saline (6%) will increase the volume of sputum expectorated over a 24 hour period compared to nebulised isotonic saline (0.9%) in patients with mild to severe stable bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* Non CF Bronchiectasis
* 18-80 years
* FEV1 less than 90%
* Chronic sputum production
* Clinical stable

Exclusion Criteria:

* Intolerance to HTS
* Use of HTSaline or antibiotics 14 days prior to study
* Clinically unstable
* Smokers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
24 hour sputum volume | 13 weeks
  24 hour volume sputum

SECONDARY OUTCOMES:
Pulmonary Function Testing | 13 weeks
  Spirometry (FEV1 and FVC) will assess the side effects using HTS.
Rheology | 13 weeks
  Rheology is the measurement of the viscosity and elasticity of sputum (viscoelasticity) and also the thread forming ability of mucus (spinnibility). Rheology will assess the extent to which HTS effect the viscosity of secretions and rehydrates secretions by drawing water into the mucus via osmosis.
Adherence | 13 weeks
  All used and unused vials of the study drug shall be counted. The researcher will review the returned vials (used and unused) along with the patient diary cards, which record information regarding airway clearance and administration of study drug.
Patient Reported Outcomes RSSQ | 13 weeks
  RSSQ: a signs and symptoms questionnaire used in clinical trials in order to diagnose an exacerbation.
Patient Reported Outcome: Leicester Cough Questionnaire: | 13 weeks
  Leicester Cough Questionnaire: a valid and reliable health status measure for adults with chronic cough
  Quality of Life Questionnaire Bronchiectasis (QOL-B), a tool used to evaluate quality of life in patients with bronchiectasis.
Bronchiectasis Qol Questionnaire | 13 weeks
  Bronchiectasis Qol Questionnaire is a disease specific questionnaire developed to assess disease specific QOL in Bronchiectasis

CONTACTS AND LOCATIONS:
Locations (1):
- Belfast HSCT, Belfast, Northern Ireland, United Kingdom